CLINICAL TRIAL: NCT01293903
Title: A Multi-center, Randomized, Double, Placebo-controlled, Parallel Group Study of Improving Heart Function and Immunoregulation Effects of Qiliqiangxin Capsule in Patients With Dilated Cardiomyopathy
Brief Title: Study of Qiliqiangxin Capsule to Treat Dilated Cardiomyopathy
Acronym: QLQX-DCM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Fudan University (Other); First Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Shandong Provincial Hospital (Other Government); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Ministry of Science and Technology of the People´s Republic of China (Other Government); China National Center for Cardiovascular Diseases (Other Government); RenJi Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); Wuhan University (Other); Henan Provincial People's Hospital (Other); Jining Medical University (Other); Second Hospital of Shanxi Medical University (Other); Shanxi Cardiovascular Hospital (Other); Wuhan Pu-Ai Hospital (Other); Tianyou Hospital Affiliated to Wuhan University of Science and Technology (Other); Yunyang Medical College (Other); China Three Gorges University, Yichang, China (Other); Xiangyang Central Hospital (Other); Wuhan No.1 Hospital (Other); Jingzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hua Liao, Professor and director of Institute of Cardiology, Union Hospital, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLQX-DCM-01
Record Dates: First submitted 2011-01-31; First posted 2011-02-11 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Dilated Cardiomyopathy; Heart Failure
Keywords: Immunomodulation
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure | interventions — qiliqiangxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qiliqiangxin capsule (Experimental)
  Interventions: Drug: Qiliqiangxin capsule
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qiliqiangxin capsule — Qiliqiangxin capsule is administrated based on the standard heart failure treatment in China. Dosage: 1.2g/times. Frequency: 3 times/day. Duration: The whole study period.
  Arms: Qiliqiangxin capsule
Drug: Placebo — Placebo, similar in color and taste to Qiliqiangxin capsule, is administrated based on the standard heart failure treatment in China. Dosage: 1.2g/times. Frequency: 3 times/day. Duration: The whole study period.
  Arms: Placebo

SUMMARY:
The pathogenesis of dilated cardiomyopathy (DCM) leading to heart failure is closely associated with autoimmunity dysfunction. A few studies represented that Qiliqiangxin capsule, a Chinese medicine, could enhance heart function in chronic heart failure and regulate the balance of TNF-a and IL-10 in myocardial infarction. In this study, to explore the effects of Qiliqiangxin capsule on the improving heart function and immunoregulation in patients with DCM, patients were recruited, anti-heart autoantibodies and some representative cytokines were assayed by enzyme-linked immuno sorbent assay (ELISA), and the efficacy of heart function improvement was compared between Qiliqiangxin capsule and placebo under the standard treatment of DCM.

ELIGIBILITY:
Inclusion Criteria:

* Dilated Cardiomyopathy (LVEF ≤ 45%)

Exclusion Criteria:

* Secondary dilated cardiomyopathy (such as ischemic cardiomyopathy, valvular cardiomyopathy, hyperthyroid cardiomyopathy, diabetic cardiomyopathy, anemia cardiomyopathy, and etc.)
* Coronary heart disease
* Rheumatic heart disease
* Pulmonary heart disease
* Continuous dysarteriotony: hypertension(systolic blood pressure [SBP] ≥ 60mmHg/diastolic blood pressure [DBP] ≥ 100mmHg); hypotension(SBP < 90mmHg/DBP < 60mmHg)
* Resting heart rate ≤ 50bpm
* Atrioventricular block patients without permanent pacemaker

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12-31 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
The value of left ventricular end-diastolic dimension (LVEDd) and left ventricular ejection fraction(LVEF) confirmed by ultrasonic cardiogram (UCG) | 12 months after intervention
The levels of serum representative cytokines detected by ELISA | 12 months after intervention

SECONDARY OUTCOMES:
Heart failure aggravation | 12 months after intervention
All cause mortality | 12 months after intervention
Sudden cardiac death | 12 months after intervention
Stroke | 12 months after intervention
The dynamic changes of serum representative cytokines detected by ELISA in the treatment group | 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hua Liao, Docter, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Tang H, Zhong Y, Zhu Y, Zhao F, Cui X, Wang Z. Low responder T cell susceptibility to the suppressive function of regulatory T cells in patients with dilated cardiomyopathy. Heart. 2010 May;96(10):765-71. doi: 10.1136/hrt.2009.184945. PMID 20448127
- [Background] Yuan J, Yu M, Lin QW, Cao AL, Yu X, Dong JH, Wang JP, Zhang JH, Wang M, Guo HP, Cheng X, Liao YH. Th17 cells contribute to viral replication in coxsackievirus B3-induced acute viral myocarditis. J Immunol. 2010 Oct 1;185(7):4004-10. doi: 10.4049/jimmunol.1001718. Epub 2010 Aug 27. PMID 20802148
- [Background] Xiao H, Wang M, Du Y, Yuan J, Cheng X, Chen Z, Zou A, Wei F, Zhao G, Liao YH. Arrhythmogenic autoantibodies against calcium channel lead to sudden death in idiopathic dilated cardiomyopathy. Eur J Heart Fail. 2011 Mar;13(3):264-70. doi: 10.1093/eurjhf/hfq198. Epub 2010 Nov 2. PMID 21044990
- [Background] Xiao H, Song Y, Li Y, Liao YH, Chen J. Qiliqiangxin regulates the balance between tumor necrosis factor-alpha and interleukin-10 and improves cardiac function in rats with myocardial infarction. Cell Immunol. 2009;260(1):51-5. doi: 10.1016/j.cellimm.2009.09.001. Epub 2009 Sep 11. PMID 19833326